CLINICAL TRIAL: NCT04724070
Title: Comprehensive Precision Oncology Program at The Chinese University of Hong Kong
Brief Title: PRecision Oncology CUhk pRogrammE (PRO-CURE)
Status: Recruiting | Type: Observational
Sponsor: Brigette Ma (Other)
Responsible Party: Sponsor-Investigator, Brigette Ma, Professor, Department of Clinical Oncology, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Other Study IDs: PROCURE
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Gastrointestinal Cancers
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NGS and PDO/PDX establishment
  Interventions: Genetic: NGS, PDO/PDX establishment

INTERVENTIONS:
Genetic: NGS, PDO/PDX establishment — Patients' tumor specimens will be collected for next generation sequencing, PDO/PDX establishment and tissue banking.

SUMMARY:
The main aim of this project is to establish an innovative model of a comprehensive precision oncology platform to help individualizing drug therapy for patients with advanced cancers at The Chinese University of Hong Kong. The other objectives include to optimize the genomic matching and access of patients with unique cancer subtypes to the relevant clinical trials of novel therapies, and to construct a personalized drug screening platform for individuals using novel cancer models established from patient-derived cancer cells and tissues. Other objectives include to investigate the utility and feasibility of genomic sequencing using circulating tumor DNA(ctDNA), and to establish a biobank of tumor tissues derived from patients with unique cancer subtypes.

ELIGIBILITY:
Inclusion Criteria:

* Must be aged between 18 to 75 years
* Must have ECOG performance status of 0 to 1
* Must have histologically/cytologically confirmed cancers of certain subtype
* Medically fit patients who would need systemic therapy as part of their oncological treatment in any one or more of the following oncological setting(s): palliative, neoadjuvant, adjuvant, concurrent with radiotherapy. This includes patients who have limited systemic therapeutic options for their cancers and are candidates for clinical trials.
* Able to give written informed consent
* Willing to have blood samples taken.
* Availability of an archived paraffin-embedded tumor block

Exclusion Criteria:

* Patients who refuse or are medically unfit for systemic therapy for their cancer
* Patients with more than one invasive cancers diagnosed over the last FIVE years.
* Patients without measurable tumor lesions on radiological imaging
* Patients who are unable to give written informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cancer types that are allowed in this study:
  * Gastrointestinal cancers: esophageal cancer, colorectal cancer, gastric cancer, esophago-gastric junction cancer, pancreatic cancer (including neuroendocrine cancers), small bowel cancer, appendiceal cancer, anal cancer.
  * Cancers that are known to carry unique genomic aberrations that are clinically relevant and/or potentially actionable.
  Excluded types of neoplastic or dysplastic disorders:
  - Lymphoma, leukemia, lymphoproliferative disease, plasma cell neoplasms, histiocytosis-related proliferative disorders.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-10-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Establishment of an innovative model of a comprehensive precision oncology platform | 4 years
Construction of a personalized drug screening platform for individuals using novel cancer models established from patient-derived cancer cells and tissues. | 4 years

SECONDARY OUTCOMES:
Describe the prevalence of actionable genomic aberrations in patients with advanced cancers in Hong Kong | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No